CLINICAL TRIAL: NCT04052685
Title: Selective Removal to Soft Dentine or Selective Removal to Firm Dentine for Deep Caries Lesions in Permanent Posterior Teeth: A Randomized Controlled Trial up to 5 Years
Brief Title: Selective Removal to Soft Dentine vs Selective Removal to Firm Dentine for Deep Posterior Caries Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: burcu gözetici (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor-Investigator, burcu gözetici, Asst. Prof., Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.53565
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Deep Caries; Pulp Exposure, Dental; Dental Caries
MeSH Terms: conditions — Dental Pulp Exposure; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective removal to soft dentin (SRSD) (Experimental): The patients in SRSD group will be randomized into two subgroups as Group A and Group C. After caries removal to soft dentin calcium silicate based material (Biodentine) will be applied in Group A while will not be applied in Group C prior to placement of the resin composite restoration. The procedure, starts with access to caries tissue by the removal of surrounding unsupported enamel.Carious tissue at the periphery of the cavity will be prepared to hard dentin using round tungsten carbide burs and/or an excavator, while soft carious dentin will remain in the pulpal aspect of the cavity to prevent pulp exposure. Operative procedures will be performed by an experienced (over 10 years) specialist. Moisture control will be provided using cotton rolls and continuous aspiration.
  Interventions: Procedure: Selective removal to soft dentin (SRSD)
- Selective removal to firm dentin (SRSD) (Active Comparator): Procedures will be done using local anesthesia. The procedure, starts with access to caries tissue by the removal of surrounding unsupported enamel. Caries tissue in the periphery including the enamel-dentinal junction will be removed using round tungsten carbide burs and/or an excavator until hard, dry dentin remains. Pulpo-proximal caries tissue will be removed until hard or leathery dentin remains. Operative procedures will be performed by an experienced (over 10 years) specialist. Moisture control will be provided using cotton rolls and continuous aspiration. Restoration will be performed after caries removal to firm dentin and placement of calcium silicate based material (Biodentine).
  Interventions: Procedure: Selective removal to firm dentine (SRFD)

INTERVENTIONS:
Procedure: Selective removal to soft dentin (SRSD) — In order to prevent pulp exposure in deep caries lesions radiographically extending at least 3/4 of dentin, periphery of the cavity prepared to hard dentin while reasonable amount of soft carious tissue over the pulp is left. This caries removal strategy is termed selective removal to soft dentine.
  Other Names: Partial caries excavation; Incomplete caries excavation
  Arms: Selective removal to soft dentin (SRSD)
Procedure: Selective removal to firm dentine (SRFD) — Carious tissue is totally removed until hard dentin dry in appearance and hard on probing. This carious removal strategy is strongly recommended for shallow or moderately deep carious lesions.
  Other Names: Total caries removal
  Arms: Selective removal to firm dentin (SRSD)

SUMMARY:
Removal of infected dentin contaminated with bacteria and remaining affected dentin detected as firm is the conventional strategy for the management of cavitated caries lesions. Recently, this strategy is termed as selective removal to firm dentin (SRFD) and seems to increase the potential risk of pulp exposure or loss of pulp vitality for deep caries lesions radiographically extending ¾ of dentin tissue. Alternatively, selective removal to soft dentine (SRSD) that refers to removal of caries tissue at the periphery of the cavity to firm dentin and remaining caries tissue detected as soft or leathery in proximity with the pulp might be a less invasive excavation method for deep caries lesions to maintain pulpal health. However, information on clinical advantages or disadvantages of SRSD and SRFD excavation methods is sparse and mostly rely on studies conducted for primary teeth. Moreover, clinical trials are needed to demonstrate the combined effect of carious removal strategies and calcium silicate-based materials.

The aim of this study is comparison of clinical success rates of SRSD and SRFD techniques in posterior deep caries lesions. The primary outcome of the study is comparison of clinical success of SRSD and SRFD techniques by clinical and radiographic examination after 3 months, 6 months, 1 year and 2 years. The secondary outcome of the study is to investigate whether or not calcium silicate-based materials have an effect on the success rate of the treatment.

DETAILED DESCRIPTION:
In recent years, there has been growing number of studies questioning conventional caries tissue removal, especially for deep caries lesions (1). In the concept of conventional caries tissue removal, 'affected dentin' and 'infected dentine' are widely used terms which have been defined by Massler (2) in 1960s. According to this concept, removal of infected dentin contaminated with bacteria and remaining affected dentin detected as firm suggested for the management of cavitated caries lesions. Recently, this removal technique is termed as selective removal to firm dentin (SRFD) and seems to increase the potential risk of pulp exposure or loss of pulp vitality for deep caries lesions radiographically extending ¾ of dentin tissue (3). In case of pulp exposure, direct pulp capping is the treatment of choice for a tooth with a vital pulp and without any inflammation predictors such as prolonged bleeding. However, according to results of a long term (5-10 years) retrospective study evaluating the treatment outcome of direct pulp capping with calcium hydroxide, 44.5% in the 5-yr group and 79.9% in the 10-yr group had a postoperative root canal treatment or an extraction (4). Similarly, another restrospective study showed that over the first year after direct pulp capping with calcium hydroxide , almost 10% and, after 5 years, nearly 20% of the teeth had an unfavourable treatment outcome (5).According to results of these studies, survival rate of directly capped pulp tissue with calcium hydroxide seems to decrease over time.

Recently, Biodentine (BD; Septodont, St Maur-des-Fosses, France), which is a calcium silicate-based material, has gained popularity for pulp capping treatment. The success rate of Biodentine reported to be 91.7% after 3 years in a recent prospective longitudinal randomized controlled study of vital permanent teeth with deep caries (6). Except from the material of choice for pulp capping, some other strategies such as selective removal to soft dentin (SRSD) has been recently recommended for the management of deep caries lesions with the aim of reducing the risk of pulp exposure.

Accorging to report of International CariesConsensus Collaboration (ICCC) group SRSD is strongly recommended in deep cavitated lesions extending into ¾ of dentin tissue. Soft carious tissue is left over the pulp to avoid pulpal exposure and peripheral enamel and dentine are prepared to hard dentine, to provide hermetic sealing and durability of the restoration.

In the literature, there are very few studies concerned with the clinical success of SRSD, incomplete caries removal (ICR) or partial caries removal (PCR). In a long term (10 years) prospective cinical study, the success rates of PCR technique has been reported as, 90% after 3 years, 82% after 5 years and %63 after 10 years (7). In another clinical study comparing 24-month pulp health outcomes of PCR and total caries removal (TCR) in primary molars, no significant diffrence between the two removal techninues and reduced risk for pulp exposure with PCR technique has been reported (8). In a recently published review, it has been reported that SRSD seems to be the best option for the treatment of deep caries lesions and the remaining caries tissue close to the pulp seems not to interfere the longevity of the restorations (9).Nevertheless, not much scientific evidence on clinical success of SRSD and SRFD excavation methods for deep carious lesions in permanent teeth could be found in the currently available literature. Moreover, clinical trials are needed to demonstrate the combined effect of carious removal strategies and calcium silicate-based materials.

The aim of this study is comparison of clinical success rates of SRSD and SRFD techniques in posterior deep caries lesions of permanent teeth. This study will be carried out as a prospective randomized, double-blinded, clinical trial, with 2 parallel groups. Potential patients attending to Istanbul Medipol University Dental Clinics in Istanbul with deep posterior caries lesions will be invited to the study. The patients meeting the inclusion criteria will be recruited and randomized into SRSD group and SRFD group by block randomization of 2.1 ratio.

After giving their consent to take part in the study, defined clinical procedure for each group will be performed. In SRFD group (Goup B), after caries removal to firm dentin calcium silicate based material (Biodentine) will be applied. If the excavations led to pulp exposure, pulp-capping with calcium silicate based material will be performed and this patients will be randomized to another group (Group PC).The patients in SRSD group will be randomized into two subgroups as Group A and Group C. In group A after caries removal to soft dentin calcium silicate based material (Biodentine) will be applied. In group C after caries removal universal adhesive material will be applied without calcium silicate based material placement. All the restorations will be performed by the same operator using the same universal adhesive and resin composite material. The observers (two independent observer) and the patients will be blinded for the actual intervention performed.

The primary outcome of the study is comparison of clinical success of SRSD and SRFD techniques by clinical and radiographic examination after 3 months, 6 months, 1 year and 2 years. The secondary outcome of the study is to investigate whether or not calcium silicate-based materials have an effect on the success rate of the treatment. Statistical comparisons will be performed between Group A and Group B for the primary outcome and between Group A and Group C for the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Deep primary active caries lesion extending at least 3/4 of dentin
* No irreversible pulpitis symptoms
* Positive response to electrical and cold pulp vitality tests
* Good general health
* No untreated periodontal disease
* Acceptance to be included in study

Exclusion Criteria:

* Irreversible pulpitis symptoms
* Negative response to electrical and cold pulp vitality tests
* Radiographically periradicular pathology
* Pregnancy
* Teeth with non-carious lesions (attrition, erosion, abrasion or abfraction)
* Patients planning bleaching or orthodontic treatment
* Known allergy to study material

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Success (endodontic treatment required no/yes) | 60 months
  The primary outcome of the study will be success (i. e. not requiring root canal treatment intervention).
  Pulp vitality (yes/no), pain on percussion or palpation (yes/no), presence of abscess or fistula (yes/no) will assessed clinically. Radiographically, periradicular pathology (yes/no), pathologic calcification or resorption (yes/no) will be assessed.
Post-operative sensitivity (yes/no) | 60 months
  The second outcome of the study will depend on Patients' subjective assessment of the treatment (severe/moderate/no)

SECONDARY OUTCOMES:
Dentin bridge formation | 60 months
  Whether or not placement of calcium silicate based material (Biodentine) has an extra benefit for dentin bridge formation (dentin bridge formation yes/no)
Restoration integrity | 60 months
  Restorations will be evaluated according to FDI World Dental Federation criteria (10). This instrument is composed of three dimensions (biological, functional and esthetic). Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome (1:excellent; 2:clinically good; 3:clinically satisfactory; 4:unsatisfactory but repairable; 5: replacement necessary).
  Esthetic Properties:
  * Surface Luster (1-5)
  * Staining (1-5)
  * Color match and translucency (1-5)
  * Anatomical form (1-5)
  Functional Properties:
  * Fracture of material and retention (1-5)
  * Marginal adaptation (1-5)
  * Occlusal wear (1-5)
  * Approximal anatomical form (1-5)
  * Radiographic examination (1-5)
  * Patient's view (1-5)
  Biological Properties
  * Recurrence of caries (1-5)
  * Tooth integrity (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Gözetici Çil, DDS, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Schwendicke F, Frencken JE, Bjorndal L, Maltz M, Manton DJ, Ricketts D, Van Landuyt K, Banerjee A, Campus G, Domejean S, Fontana M, Leal S, Lo E, Machiulskiene V, Schulte A, Splieth C, Zandona AF, Innes NP. Managing Carious Lesions: Consensus Recommendations on Carious Tissue Removal. Adv Dent Res. 2016 May;28(2):58-67. doi: 10.1177/0022034516639271. PMID 27099358
- [Background] Massler M. Pulpal reactions to dental caries. Int Dent J. 1967 Jun;17(2):441-60. No abstract available. PMID 5233875
- [Background] Ricketts D, Innes N, Schwendicke F. Selective Removal of Carious Tissue. Monogr Oral Sci. 2018;27:82-91. doi: 10.1159/000487838. Epub 2018 May 24. PMID 29794475
- [Background] Barthel CR, Rosenkranz B, Leuenberg A, Roulet JF. Pulp capping of carious exposures: treatment outcome after 5 and 10 years: a retrospective study. J Endod. 2000 Sep;26(9):525-8. doi: 10.1097/00004770-200009000-00010. PMID 11199794
- [Background] Dammaschke T, Leidinger J, Schafer E. Long-term evaluation of direct pulp capping--treatment outcomes over an average period of 6.1 years. Clin Oral Investig. 2010 Oct;14(5):559-67. doi: 10.1007/s00784-009-0326-9. Epub 2009 Aug 15. PMID 19685086
- [Background] Awawdeh L, Al-Qudah A, Hamouri H, Chakra RJ. Outcomes of Vital Pulp Therapy Using Mineral Trioxide Aggregate or Biodentine: A Prospective Randomized Clinical Trial. J Endod. 2018 Nov;44(11):1603-1609. doi: 10.1016/j.joen.2018.08.004. Epub 2018 Oct 3. PMID 30292451
- [Background] Maltz M, Alves LS, Jardim JJ, Moura Mdos S, de Oliveira EF. Incomplete caries removal in deep lesions: a 10-year prospective study. Am J Dent. 2011 Aug;24(4):211-4. PMID 22016914
- [Background] Franzon R, Guimaraes LF, Magalhaes CE, Haas AN, Araujo FB. Outcomes of one-step incomplete and complete excavation in primary teeth: a 24-month randomized controlled trial. Caries Res. 2014;48(5):376-83. doi: 10.1159/000357628. Epub 2014 Apr 8. PMID 24732081
- [Background] Carvalho JC, Dige I, Machiulskiene V, Qvist V, Bakhshandeh A, Fatturi-Parolo C, Maltz M. Occlusal Caries: Biological Approach for Its Diagnosis and Management. Caries Res. 2016;50(6):527-542. doi: 10.1159/000448662. Epub 2016 Sep 23. PMID 27658123
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation - clinical criteria for the evaluation of direct and indirect restorations. Update and clinical examples. J Adhes Dent. 2010 Aug;12(4):259-72. doi: 10.3290/j.jad.a19262. PMID 20847997
- [Derived] Gozetici-Cil B, Erdem-Hepsenoglu Y, Tekin A, Ozcan M. Selective removal to soft dentine or selective removal to firm dentine for deep caries lesions in permanent posterior teeth: a randomized controlled clinical trial up to 2 years. Clin Oral Investig. 2023 May;27(5):2125-2137. doi: 10.1007/s00784-022-04815-0. Epub 2022 Dec 3. PMID 36460919